CLINICAL TRIAL: NCT02131961
Title: A Study to Evaluate the Feasibility of Using a Modified Cast Walker With a Portal for Application of Topical Medications in Diabetic Foot Ulcers
Brief Title: EZCast-DFU Study With Portal for Application of Topical Medications
Acronym: EZCast-DFU
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Robert S. Kirsner, Professor, Vice Chairman Department of Dermatology & Cutaneous Surgery, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20140171
Record Dates: First submitted 2014-05-02; First posted 2014-05-06 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Foot Ulcer; Diabetic Foot
Keywords: diabetic foot; foot ulcer; foot wound; plantar ulcer; plantar wound; contact cast; collagenase
MeSH Terms: conditions — Foot Ulcer; Diabetic Foot; Foot Injuries | interventions — Collagenases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study arm (Experimental): Collagenase ointment topical application, once daily for 14 days, modified Contact Cast System, applied at days 0,3, and 7.
  Interventions: Drug: Collagenase ointment; Device: Modified Contact Cast System

INTERVENTIONS:
Drug: Collagenase ointment — 250 collagenase units/g
  Other Names: Santyl
Device: Modified Contact Cast System — 1 Unit
  Other Names: Modified TCC-EZ(R) Total Contact Cast System

SUMMARY:
This study is designed to evaluate the ability to modify a contact cast system so that topical medications can be applied daily to an underlying wound in patients with diabetic plantar ulcers. The modification of the cast will be done by making an opening where the wound is located in the contact cast system. A contact cast system is a device that will reduce the pressure in the area where the wound is located.

DETAILED DESCRIPTION:
The accepted care of a diabetic foot ulcer includes cleaning of the wound of the dead and dying tissue around the wound, daily wound care, good nutrition, and adequate relief of pressure. Pressure reduction, commonly known as "off-loading," is most often achieved by having the patient wear an "off-loading boot". However, using a cast similar to the cast used to treat broken bones will result in less activity and better wound healing. The cast is considered the best method for off-loading the foot but is not used as often as other methods because the cast covers the foot ulcer and it does not allow you to perform daily cleaning and examination.

This study will apply a Total Contact Cast (TCC)System and leave an opening where the ulcer can be treated on a daily basis by the investigators. Patients will be asked to apply an ointment called Santyl ® to their ulcer on a daily basis. Santyl ® ointment is an FDA approved drug that is routinely used on foot ulcers. The Santyl ® ointment cleans wounds to promote a better environment for wounds to heal. It helps remove nonliving tissue without harming the new healing tissue.

Trial will last 14 days and it will consist of 4 visits. In the first visits, patients' wounds will be cleaned from dead and dying tissue (debridement) and the first modified contact cast will be applied. Patients will be provided Santyl to apply daily with reapplication of foam dressing. Patients will return at day 3, and then weekly for 2 weeks for standard evaluation and debridement and wound measurements and at day 3, and week 1 visit for reapplication of the modified contact cast.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 18 and 80 years of age (inclusive) with diabetes type 1 or type 2
* Patients must sign an informed consent
* Diabetic medications must be stable for 4 weeks prior to randomization.
* Patients with a plantar ulcer
* Ulcer with an area between ≥ 1 cm2 and ≤ 10 cm2
* Patients must agree to comply with at least daily dressing changes and off-loading according to protocol requirements;
* Ulcer at least 6 weeks but not more than 12 months old
* Diabetic patients who use a medication to lower blood glucose levels who, in the opinion of the investigator, are considered "controlled" diabetics
* Adequate perfusion of the foot with the ulcer
* No prior use of Santyl on the target ulcer or treatment within one month with other bioactive therapies

Exclusion Criteria:

* Patients with more than two ulcers on the same foot
* Patients with ulcer requiring off-loading that cannot be effectively off-loaded
* Patients with ulcer above the plantar foot;
* Patient non-compliance with protocol-required off-loading and dressing change
* Patients with infected ulcers
* Patients with severe edema (defined as inability to fit leg into off-loading device);
* Patients with a gangrenous or ischemic toe that may need to be amputated in the opinion of the investigator;
* Patients with Buerger's disease, vasculitis or connective tissue disease;
* Ankle brachial index >1.2 (ABI >1.2 must be confirmed by another method such as Transcutaneous partial pressure oxygen (TcPO2) > 40 mm Hg at the ankle or Toe pressure of > 40mm Hg or Doppler waveform consistent with adequate flow in the foot (biphasic or triphasic) or Skin Perfusion Pressure (SPP) > 40 mm Hg);
* Patients with claudication
* Body mass index (BMI) > 40 kg/m2
* There is active Charcot's joint by clinical or radiographic criteria.
* Unable or unwilling to provide informed consent.
* Known HIV infection and/or AIDS based on participant self-report.
* Patients with contraindication to contact casting (ie. peripheral vascular disease, Infection)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Proportion of contact cast systems intact by day 14 | 14 days
  Proportion of contact cast systems in whom the investigator assesses as intact (not damaged, or broken by the creation of the window).
  Intact: Contact cast systems where the window creation did not create unintended fissures or these fissures were less than 1cm length and they originate from the window opening.
  Damaged: Contact cast systems where window creation creates one or more fissure between 1-3cm of length and these fissures originate from the window opening.
  Broken: Contact cast systems where window creation creates one or more fissures of length more than 3 cm, or any fissure that did not originate from the site of the window opening

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Kirsner, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, University of Miami Hospital & Clinics, Miami, Florida, United States

REFERENCES:
- See also: Wound Research Clinic. University of Miami — http://dermatology.med.miami.edu/research/cutting-edge-wound-research